CLINICAL TRIAL: NCT00120341
Title: A Randomized, Double Blind, Placebo Controlled Prospective Study to Evaluate the Effectiveness of Monochromatic Infrared Photo Energy to Improve Diabetic Sensory Neuropathy
Brief Title: Anodyne Therapy in Diabetic Sensory Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Collaborators: Anodyne Therapy, LLC (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 50100
Record Dates: First submitted 2005-06-30; First posted 2005-07-15 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes Mellitus; Diabetic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies

INTERVENTIONS:
Device: Anodyne Therapy System

SUMMARY:
The purpose of this research study is to determine if the use of a series of the Anodyne Therapy System in-home treatments over a 90-day period will improve peripheral sensation and quality of life in persons with diabetes mellitus.

DETAILED DESCRIPTION:
The morbidity, direct cost and mortality associated with lower extremity complications among patients with diabetes mellitus have been well described in the medical literature. Peripheral sensory neuropathy is one of the strongest risk factors for both foot ulceration and amputation in this population. In the absence of neuropathy people rarely develop foot ulcers. Because of the lack of painful feedback, peripheral neuropathy provides a permissive environment that allows repetitive tissue injury to occur such that a person may wear a hole in the bottom of his or her foot much in the way that he or she may wear a hole in a stocking. Certainly, the early detection of a level of peripheral neuropathy sufficient to contribute to the development of foot wounds or "loss of protective sensation" is one of the most important criteria to identify high risk patients for foot complications and is paramount when instituting a structured treatment plan to prevent lower extremity complications.

The objective of the study is to determine the efficacy of the application of a series of Anodyne in-home treatments over a 90-day period to improve peripheral sensation and self-reported quality of life in persons with diabetes mellitus. This pilot study should provide preliminary data to determine if additional clinical evaluation is warranted and to determine an appropriate sample size. The hypothesis is the Anodyne therapy will improve sensory function over the course of therapy compared to sham therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetes mellitus and peripheral sensory neuropathy.
* Subjects at least 25 years old.
* Vibration perception threshold (VPT) ≥ 20 volts and ≤ 45 volts.
* Subjects must be alert, oriented, mentally competent and able to understand and comply with the requirements of the study, and provide voluntary informed consent.
* Subjects must be willing and able to complete the required study visits and record treatment activity in the study logbook.

Exclusion Criteria:

* Subjects who have a VPT <20 or > 45 volts.
* Subjects with uncontrolled hypertension greater than 180 systolic or greater than 110 diastolic as determined by enrollment questionnaire
* Subjects who are pregnant or breastfeeding or who are likely to become pregnant during the course of the study.
* Subjects with active malignancy (including basal cell carcinoma) on the lower extremities.
* Subjects who have had prior reconstructive or replacement knee surgery with neurological deficits related to the surgery. ( If the patient has had knee surgery, their neuropathy appears to be uniform and bilateral, then they can be included in the study).
* Subjects with a history of previous back surgery, spinal stenosis, or spinal compression or radiculopathy with neurological deficits related to spinal cord pathology. ( If the patient has had back surgery, their neuropathy appears to be uniform and bilateral, then they can be included in the study).
* Subjects who are non-ambulatory.
* Subjects with a history of neuromuscular disease, leprosy, chronic alcoholism, or sarcoidosis.
* Subjects with foot ulcerations.
* Subjects with a transmetatarsal amputation or higher

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-04; Study Completion 2006-06

PRIMARY OUTCOMES:
changes in sensation using, vibration perception threshold testing, monofilament testing, and the Michigan Neuropathy Screening Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, Principal Investigator — Scott and White Memorial Hospital & Clinic
Locations (1):
- Scott and White Santa Fe Center, Temple, Texas, United States

REFERENCES:
- [Derived] Lavery LA, Murdoch DP, Williams J, Lavery DC. Does anodyne light therapy improve peripheral neuropathy in diabetes? A double-blind, sham-controlled, randomized trial to evaluate monochromatic infrared photoenergy. Diabetes Care. 2008 Feb;31(2):316-21. doi: 10.2337/dc07-1794. Epub 2007 Oct 31. PMID 17977931